CLINICAL TRIAL: NCT06231511
Title: Soft Exosuits for Functional Gait Recovery in Acute Stroke Rehabilitation
Status: Completed | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Director, Max Nader Center for Rehabilitation Technologies & Outcomes Research, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00210500
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Acute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (3):
- AIM 1: Single Group (Hip Flexion Soft Exosuit) (Experimental): For AIM 1, all participants are assigned to the training group using a hip flexion soft exosuit. During the training/tuning sessions, individuals will perform up to 60 minutes of walking with the exosuit on the treadmill, overground or completing stairs, with rest breaks as needed. Goals during these sessions are to modify and update the controllers for the exosuit to appropriately provide assistance to the patient while ambulating in collaboration with Harvard University. We may also test clinical training progressions with the exosuit during walking training. Some part of the session may include walking with the exosuit assisting and other part of the session may include without the device assisting for comparison. Total session time for each session may be up to 2 hours, and up to 8 training/tuning visits will be performed.
  Interventions: Device: Hip flexion soft exosuit
- AIM 2: Device Group (ReWalk ReStore Soft Exosuit) (Experimental): For participants in the experimental group, these exosuits will be utilized in up to all physical therapy sessions during the course of the patient's inpatient stay. With the consideration that an inpatient stay may be up to 10 weeks, total number of sessions may be up to 75 visits. Sessions will vary from 30-90 minutes depending on inpatient therapy scheduling.
  Interventions: Device: ReWalk ReStore soft exosuit
- AIM 2: Control Group (Active Comparator): Participants in the control group will participate in conventional physical therapy without use of exosuits during the course of the patient's inpatient stay. With the consideration that an inpatient stay may be up to 10 weeks, total number of sessions may be up to 75 visits. Sessions will vary from 30-90 minutes depending on inpatient therapy scheduling.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Device: Hip flexion soft exosuit — Participants will utilize a Wyss designed hip flexion soft exosuit. This device has a small rope winch at the front of the hip connected to a functional textile waistband and thigh band. It applies an assistive torque in response to wearable sensor measurements.
  Arms: AIM 1: Single Group (Hip Flexion Soft Exosuit)
Device: ReWalk ReStore soft exosuit — Participants will utilize the ReWalk ReStore ankle soft exosuit. This device provides dynamic plantarflexion and dorsiflexion during walking intended to restore paretic limb function resulting in improved gait symmetry, reduced energy cost of walking and improved stability. The exosuits consists of a body-worn actuation unit containing motors, gears, and pulleys that when powered generate forces that are transmitted via Bowden cables to functional textiles anchored proximal and distal to a joint. This actuation occurs in response to signals from embedded wearable sensors.
  Arms: AIM 2: Device Group (ReWalk ReStore Soft Exosuit)
Other: Conventional physical therapy — Participants will complete conventional physical therapy without use of exosuits during the course of their inpatient rehabilitation stay.
  Arms: AIM 2: Control Group

SUMMARY:
The purpose of this study is to develop and evaluate the use of soft exosuits in patients post stroke.

DETAILED DESCRIPTION:
AIM 1: Develop individualized adaptive controller parameters and a training progression program for these exosuits specific for inpatient stroke rehabilitation.

AIM 2: Evaluate the impact of the soft exosuit + conventional inpatient rehabilitation vs.

conventional inpatient rehabilitation alone on measures of lower-extremity impairments and functional recovery following acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years
* History of single stroke event with deficits predominately affecting one side of the body
* Stroke less than 4 years ago (AIM 1)
* Stroke within the past 6 months (AIM 2)
* Capable of standing with assistance
* Medical clearance by a physician

Exclusion Criteria:

* Inability to communicate with investigators
* Pressure ulcers or skin wounds located where the exosuit interfaces (calf, thigh, waist)
* History of significant peripheral artery disease (PAD)
* Unresolved deep vein thrombosis (DVT)
* Psychiatric or cognitive impairments that may interfere with proper operation of the device
* Known urethane allergies
* Pregnancy
* Other comorbidities that prevent full participation in research

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AIM 1: Single Group (Hip Flexion Soft Exosuit) | AIM 2: Device Group (ReWalk ReStore Soft Exosuit) | AIM 2: Control Group
Started | 15 | 6 | 5
Completed | 14 | 5 | 5
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIM 1: Single Group (Hip Flexion Soft Exosuit) | AIM 2: Device Group (ReWalk ReStore Soft Exosuit) | AIM 2: Control Group | Total
Number analyzed (Participants) | 14 | 5 | 5 | 24
Age, Continuous [Mean (Full Range); unit: Years] | 56.7 [37 to 72] | 54.0 [37 to 69] | 54.8 [42 to 70] | 55.8 [37 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 3 | 13
  Male | 8 | 1 | 2 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 1 | 7
  White | 10 | 3 | 4 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 5 | 5 | 24
10 Meter Walk Test [Mean (Full Range); unit: m/sec] | 0.22 [0.05 to 0.72] | 0.30 [0 to 0.67] | 0.46 [0.17 to 0.75] | 0.28 [0 to 0.75]

OUTCOME MEASURES:

1. Primary Outcome: Change in 10 Meter Walk Test
Description: This test will examine the patient's gait speed. Patients will be directed to walk at their preferred and maximum but safe speed. Patients will be positioned 1 meter before the start line and instructed to walk the entire distance and past the end line approximately 1 meter. The distance before and after the course are meant to minimize the effect of acceleration and deceleration. Time will be recorded using a stopwatch and recorded to the one hundredth of a second (ex: 2.15 sec). The data table shows the change in gait speed (meters per second) from admission to discharge, time frame varies based on length of stay (estimated 2-4 weeks).
Time Frame: Admission time-point to discharge time-point (estimated 2-4 weeks). Pre-assessment completed after admission to inpatient rehabilitation, prior to first intervention session. Post-assessment completed following last treatment session, prior to discharge.
Measure: Mean (Full Range); unit: m/sec
Arm/Group | AIM 1: Single Group (Hip Flexion Soft Exosuit) | AIM 2: Device Group (ReWalk ReStore Soft Exosuit) | AIM 2: Control Group
Number analyzed (Participants) | 14 | 5 | 5
m/sec | 0.48 [0.09 to 1.03] | 0.53 [0.14 to 1.11] | 0.78 [0.32 to 1.06]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at the beginning of each session, up to 7 sessions, until discharge assessment was completed (estimated 2-4 weeks from admission time point, varied based on length of stay in inpatient rehabilitation)
Arm/Group | AIM 1: Single Group (Hip Flexion Soft Exosuit) | AIM 2: Device Group (ReWalk ReStore Soft Exosuit) | AIM 2: Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/15 | 2/6 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AIM 1: Single Group (Hip Flexion Soft Exosuit) (N=15) | AIM 2: Device Group (ReWalk ReStore Soft Exosuit) (N=6) | AIM 2: Control Group (N=5)
Leave of Absence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Fall Outside Study Procedures (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT06231511/Prot_001.pdf
  • Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT06231511/SAP_002.pdf
  • Informed Consent Form (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT06231511/ICF_003.pdf